CLINICAL TRIAL: NCT02903992
Title: SArcopenia Prevalence in Frail Older Adults: SAF Study
Brief Title: SArcopenia Prevalence in Frail Older Adults. SAF Study
Acronym: SAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/15/7817; 2016-A00181-50 (Other: ID-RCB)
Record Dates: First submitted 2016-06-29; First posted 2016-09-16 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Aging
Keywords: Frail Elderly; sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients recruited (Other): All patients who are enrolled in study with at least one Fried criteria will have a Dual-energy X-ray absorptiometry (DXA) to measure lean muscle mass adjusted for body mass index. As part of the usual care in the Frailty Clinic patients will also have a clinical examination, a standard biological sample (requiring 15 ml of blood); an evaluation of the cognitive and functional performances, of their medico-economic situation and lifestyle.
  Interventions: Radiation: Dual-energy X-ray absorptiometry (DXA)

INTERVENTIONS:
Radiation: Dual-energy X-ray absorptiometry (DXA) — Patients with at least one Fried criteria will have a Dual-energy X-ray absorptiometry (DXA) to measure lean muscle mass adjusted for body mass index. As part of the usual care in the Frailty Clinic patients will also have a clinical examination, a standard biological sample (requiring 15 ml of blood); an evaluation of the cognitive and functional performances, of their medico-economic situation and lifestyle.

SUMMARY:
The age-associated loss of lean mass is a defining parameter of sarcopenia and may lead to various negative health outcomes such as impairment of physical performance and disability. Furthermore sarcopenia is considered to be one of the main factors in the pathogenesis of the frailty syndrome. However, for clinical use and for treatment and prevention strategies, reliable diagnostic criteria and cutpoints based on clinically relevant thresholds are indispensable.

This topic has recently been addressed by the Foundation for the National Institutes of Health Sarcopenia Project which identified cutpoints for appendicular lean mass (ALM) below which older adults had a higher likelihood of clinically relevant weakness reflected by low grip strength. Moreover, a low ALM-to-body mass index (BMI) ratio (<0.789 men and <0.512 women) was found to be associated with increased likelihood for mobility impairment.

In this context, the aim of this study is to study the prevalence of sarcopenia in a sample of community-dwelling frail and pre-frail older adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 70 years and over,
* Living independently (ADL score ≥ 5/6),
* Fail or pre-frail according to Fried criteria,
* Informed written consent,
* Subjects affiliated to a social security.

Exclusion Criteria:

* Robusts patients (no Fried criteria),
* Other disorders that could interfere with the interpretation of the study (like visual or hearing impairments),
* Subjects under justice protection,
* Participation in another study at the same time.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sarcopenia Diagnostic with Dual-energy X-ray absorptiometry | one day (participation of subject)
  The primary outcome of SAF study is to assess the prevalence of sarcopenia in frail and pre-frail older adults. The primary endpoint is the sarcopenia diagnostic. In patients with at least one Fried criteria, we would like to detect the number of patient with low lean muscle mass adjusted for body mass index <0.789 for men and <0.512 for women.

SECONDARY OUTCOMES:
(SPPB) score | one day (participation of subject)
  Short Physical Performance Battery (SPPB) score
(MMSE) score | one day (participation of subject)
  Mini-Mental State Examination (MMSE) score
(MNA) score | one day (participation of subject)
  Mini Nutritional Assessment (MNA) score
(IADL) score | one day (participation of subject)
  Instrumental Activities of Daily Living (IADL) score

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand FOUGERE, MD, Ph D, Principal Investigator — oulouse University Hospital (CHU de Toulouse)
Locations (1):
- Toulouse University Hospital (CHU de Toulouse), Toulouse, France

IPD SHARING:
Plan to Share IPD: No